CLINICAL TRIAL: NCT05127785
Title: Frailty in Individuals With Advanced Heart Failure Part 2
Status: Withdrawn | Type: Observational
Why Stopped: Transitioned professional responsibilities.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elyse Peterson, Associate Professor of Clinical Occupational Therapy, University of Southern California
Other Study IDs: UP-21-00687
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Frailty
MeSH Terms: conditions — Heart Failure; Frailty | interventions — Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Medical Management: Patients deemed not candidates for advanced heart failure interventions.
- Left Ventricular Assist Device (LVAD): Recipients of a left ventricular assist device
  Interventions: Procedure: LVAD or Heart Transplant
- Heart Transplant: Recipients of a heart transplant.
  Interventions: Procedure: LVAD or Heart Transplant

INTERVENTIONS:
Procedure: LVAD or Heart Transplant — Patients undergoing advanced heart failure intervention including LVAD implantation or heart transplantation
  Groups: Heart Transplant; Left Ventricular Assist Device (LVAD)

SUMMARY:
To investigate how measures of frailty, assessed during occupational therapy (OT) evaluation and intervention impact decision for advanced heart failure (HF) therapies and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be included in this study if they were evaluated for advanced heart failure therapies at Keck Hospital from 1/1/2019-6/30/2021. This will be determined through data from the electronic medical record.

Exclusion Criteria:

* Patients who did not receive an occupational therapy evaluation prior to advanced heart failure intervention decision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with heart failure undergoing evaluation for advanced heart failure therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | 1 to 500 days
  Length of hospital stay after intervention
Rate of Readmission | 30 to 90 days
  Rate of Readmission after initial hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Peterson, OTD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- Keck Hospital of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No